CLINICAL TRIAL: NCT05770128
Title: Subserosal Laparoscopic Cholecystectomy for Safe Gall Bladder Surgery
Brief Title: Subserosal Laparoscopic Cholecystectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Hussein Ali, Ahmed Mohamed Hussein, Assiut University
Other Study IDs: cholecystectomy by laparoscpe
Record Dates: First submitted 2021-10-25; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Cholecystitis
MeSH Terms: conditions — Cholecystitis | interventions — Laparoscopes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: laparoscope — subserosal manipulation of gallbladder with laparoscope .

SUMMARY:
The aim is to study the safety and efficacy of subserosal laparoscopic cholecystectomy .

ELIGIBILITY:
Inclusion Criteria:

* Adult with age of or above 18 years.
* Diagnosis of chronic cholecystitis , symptomatic cholelithiasis

Exclusion Criteria:

* Previous operation or adhesion
* severe Acute Calculus pancreatitis
* gall bladder cancer
* Severe co-morbid conditions (uncontrolled diabetes, Hypertension, severe direct hyper bilirubinemia)
* Recurrent cases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: any patient admitted to surgical department wth age above 18 years old suffering & diagnosed of chronic cholecystitis , symptomatic cholelithiasis
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Detection of safety of subserosal laparoscopic cholecystectomy in comparison to conventional technique. | 6 months
  incidence of bleeding after subserosal laparoscopic cholecystectomy in comparison to conventional technique.